CLINICAL TRIAL: NCT01730898
Title: Lutein Absorption in Healthy Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: BL14
Record Dates: First submitted 2012-11-16; First posted 2012-11-21 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-07

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control capsule (Active Comparator): 2 capsules
  Interventions: Other: Study product containing lutein
- Experimental capsule (Experimental): 2 capsules
  Interventions: Other: Study product containing lutein

INTERVENTIONS:
Other: Study product containing lutein — delivered in capsule form
  Arms: Control capsule
Other: Study product containing lutein — delivered in capsule form
  Arms: Experimental capsule

SUMMARY:
This study will evaluate the absorption of lutein when consumed in different oil blends.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for the study if they meet all of the following inclusion criteria:

* BMI ≥ 18 and ≤ 25 kg/m2
* Between 18 and 45 years of age, inclusive
* Male or a non-pregnant, non-lactating female, nulliparous or at least 6 weeks postpartum prior to screening visit. A urine pregnancy test is required for all female subjects unless she is not of childbearing potential. If female is of childbearing potential, is practicing one of the following methods of birth control (and will continue through the duration of the study):

  * Condoms, sponge, diaphragm or intrauterine device;
  * Oral or parenteral contraceptives for 3 months prior to screening visit;
  * Vasectomized partner;
  * Total abstinence from sexual intercourse.
* If on a chronic medication, subject has been on constant dosage for at least two months prior to screening visit

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the following criteria:

* Current smoker
* Current chronic disease, including malabsorption or gastrointestinal disorders; hyperlipidemia; anemia; hemophilia; excessive bleeding; cystic fibrosis; kidney disease requiring dialysis; diabetes; active malignancy; wasting condition
* Current chronic contagious, infectious disease, such as active tuberculosis, Hepatitis B or C,or HIV
* Vegetarian, or has very selective food habits/dieting
* Average intake of alcoholic beverages greater than 2 drinks per day
* Medication or dietary supplement use to lower plasma lipids or affect lipid absorption or transport, including antibiotics
* Supplement use that contains carotenoids (multi-vitamin as an example)
* Known allergy or intolerance to any ingredient found in the study products

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Plasma lutein | baseline and 336 hours
  adjusted area under the curve at specified postprandial timepoint

SECONDARY OUTCOMES:
Plasma carotenoids | 2, 4, 6, 8, 12, 24, 48, and 336 hours
  mean concentrations at specified postprandial timepoints
Plasma lipid concentrations | baseline and 48 hours
  averaged concentrations at specified postprandial timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Williams, Study Chair — Abbott Nutrition
Locations (1):
- Biofortis Clinical Research, Addison, Illinois, United States